CLINICAL TRIAL: NCT01967537
Title: Evaluation of (68)Gallium- DOTATATE PET/CT for Detecting Primary and Metastatic Neuroendocrine Tumors
Brief Title: Evaluation of 68Gallium-DOTATATE PET/CT for Detecting Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 130193; 13-C-0193
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Neuroendocrine Tumors; Von Hippel-Lindau Syndrome; Hippel-Lindau Disease
Keywords: NET; MEN1; Von Hippel Lindau (VHL); Surgical Resection; Somatostatin Receptor Status
MeSH Terms: conditions — Neuroendocrine Tumors; von Hippel-Lindau Disease | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Gallium DOTATATE imaging (Experimental): 68Gallium DOTATATE imaging
  Interventions: Drug: 68Gallium DOTATATE; Procedure: Radio-guided surgery

INTERVENTIONS:
Drug: 68Gallium DOTATATE — Fasting is not required prior to the imaging study. An IV line with a large bore (21 gauge or more) will be placed preferably in the antecubital vein, and, with the patient supine, around 5mCi of the 68Ga-DOTATATE will be administered intravenously, followed by incubation for approximately 60 minutes. Then the patient will be positioned in a PET/CT scanner and images from the upper thighs to the base of the skull will be obtained. In patients with tumor induced osteomalacia, images from the top of the head to the toes will be obtained.
Procedure: Radio-guided surgery — Using 68Gallium DOTATATE

SUMMARY:
Background:

- Neuroendocrine tumors (NETs) are rare but have been more common over the past decade. The only treatment for NETs is surgery, but most are found when they are too advanced for surgery. Researchers are looking for the best way to find NETs earlier, so that surgery can be successful. They want to test if the study drug can be used along with imaging devices to detect NETs.

Objectives:

- To see how well a new experimental imaging agent, 68Gallium-DOTATATE, detects unknown primary and metastatic NETs in the gastrointestinal system and pancreas.

Eligibility:

- Adults over 10 years old with a suspected NET or family history of NET.

Design:

* Participants will be screened with a medical history and physical exam, and have a blood test.
* Participants will undergo three scans. For all of these, a substance is injected into their body, they lie on a table, and a machine takes images.
* A standard computed tomography (CT) scan of the chest, abdomen, and pelvis.
* An octreotide scintigraphy Single photon emission computed tomography (SPECT)/CT.
* A 68Gallium-DOTATATE positron emission tomography (PET)/CT. The study drug is injected into a vein, usually in the arm. Low-dose X-rays go through the body. For about 40 minutes a large, donut-shaped device takes images of the body. The entire session takes 90 to 120 minutes.
* Researchers will compare images from the three scans.
* Participants will have 1 follow-up visit each year for 5 years. At this visit, they will have a medical exam, blood taken, and a CT scan.

DETAILED DESCRIPTION:
Background:

* Neuroendocrine tumors (NETs) are rare malignancies occurring in the gastrointestinal tract, islets of the pancreas, lung, adrenal medulla and thyroid C-cells.
* Their incidence has increased over the last decade, with an incidence of 6 per 100,000 persons a year and they represent 0.46% of all malignancies.
* Most NETs are sporadic, but they can be part of familial cancer syndromes such as multiple endocrine neoplasia type 1 (MEN1), MEN2, and neurofibromatosis type 1 (NF1) or Von Hippel-Lindau (VHL) syndrome.
* Surgical resection remains the only curative treatment option for patients with NETs but 80% of patients are diagnosed with advanced (metastatic, locally inoperable, or recurrent) disease.
* The main prognostic factor in patients with NET is the extent of disease.
* The best imaging technique for detecting unknown primary and metastatic NETs has yet to be determined.
* NET cells express somatostatin receptors that can be targeted with radiolabeled 68Gallium-DOTATATE (Octreotate) for imaging purposes.
* The primary goal of this protocol is to determine the accuracy of a new somatostatin receptor targeted imaging technique, using 68Gallium-DOTATATE PET/CT to detect unknown primary and metastatic NETs.

Objectives:

-To determine the accuracy of 68Gallium-DOTATATE PET/CT scans in detecting unknown primary and metastatic gastrointestinal and pancreatic neuroendocrine tumors.

Eligibility:

* Patients with:

  * suspicion of NET on axial imaging (CT/magnetic resonance imaging (MRI)/fluorodeoxyglucose-positron emission tomography (FDG PET) and/or
  * biochemical evidence of NET (serum/urinary) based on elevated levels of chromogranin A, pancreatic polypeptide, neuron-specific enolase, vasoactive intestinal polypeptide, serotonin (urinary 5-HIAA), gastrin, somatostatin, catecholamines, metanephrines, calcitonin, fasting insulin, C-peptide (proinsulin), glucagon and/or
  * familial predisposition to NET in patients with multiple endocrine neoplasia type 1 (MEN1) and VHL.
* Age greater than or equal to 18 years of age.
* Patients must be willing to return to National Institutes of Health (NIH) for follow-up.

Design:

* Prospective study.
* A 68Ga-DOTATATE PET/CT scan will be done in patients with suspicious lesions, unknown primary tumor or metastatic gastrointestinal or pancreatic neuroendocrine disease found on anatomic imaging (CT/MRI) or in patients having biochemically active disease.
* Both functional and non-functional solid tumors will be included in this study. Furthermore, asymptomatic and symptomatic, sporadic and familial cases of NETs (such as Von Hippel-Lindau (VHL), MEN1) will be included.
* Demographic, clinical and pathologic data will be collected from the medical record and patient interview for each patient. Data will be stored in a computerized database.
* After their initial on-study evaluation, patients will be staged according to findings on imaging studies with respect to primary tumor site, size and metastases. Surgical resection of NET and/or medical managements will be recommended based on standard practice guidelines. In patients who undergo surgical treatment, the samples will be immediately stored until molecular analysis.
* Follow up will be done yearly for a total duration of 5 years. This includes a yearly imaging study and a biochemical and clinical evaluation, to assess tumor growth and disease progression.
* We estimate that the accrual rate will be 3-10 patients per month; the total accrual period for this study will be 10 months to 3 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with (any one of #1, #2, and/or #3):

  1. Suspicion of neuroendocrine tumors (NET) on axial imaging (computed tomography (CT)/magnetic resonance imaging (MRI)/fluorodeoxyglucose (FDG) positron emission tomography (PET) and/or
  2. biochemical evidence of neuroendocrine tumor (serum/urinary) based on elevated levels of chromogranin A, pancreatic polypeptide, neuron-specific enolase, vasoactive intestinal polypeptide, serotonin (urinary 5-HIAA), gastrin, somatostatin, catecholamines, metanephrines, calcitonin, fasting insulin, C-peptide (proinsulin), glucagon and/or
  3. familial predisposition to NET in patients with multiple endocrine neoplasia type 1 (MEN1) and Von Hippel-Lindau (VHL) (symptomatic and/or asymptomatic cases; with biochemical or anatomic imaging evidence of disease).
* Age greater than or equal to 10 years of age.
* For females: Negative urine pregnancy test OR post-menopausal for at least 2 years OR patient has had a hysterectomy.
* Patients must be willing to return to National Institutes of Health (NIH) for follow-up.
* Ability of subject or Legally Authorized Representative (LAR) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study.

EXCLUSION CRITERIA:

* Patients unwilling to undergo serial non-invasive imaging.
* Pregnant or lactating women: Pregnant women are excluded from this study because the effects of (68)Ga-DOTATATE in pregnancy are not known. Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of

  (68)Ga-DOTATATE in the mother, breastfeeding should be discontinued for at least one day if the mother receives (68)Ga-DOTATATE.
* Patients that have recognized concurrent active infection,
* Patients with the use of any investigational product or device, excluding 18F-dihydroxyphenylalanine (F-DOPA) scans, within 30 days prior to dosing.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsikitis VL, Wertheim BC, Guerrero MA. Trends of incidence and survival of gastrointestinal neuroendocrine tumors in the United States: a seer analysis. J Cancer. 2012;3:292-302. doi: 10.7150/jca.4502. Epub 2012 Jul 1. PMID 22773933
- [Background] Lawrence B, Gustafsson BI, Chan A, Svejda B, Kidd M, Modlin IM. The epidemiology of gastroenteropancreatic neuroendocrine tumors. Endocrinol Metab Clin North Am. 2011 Mar;40(1):1-18, vii. doi: 10.1016/j.ecl.2010.12.005. PMID 21349409
- [Background] Modlin IM, Lye KD, Kidd M. A 5-decade analysis of 13,715 carcinoid tumors. Cancer. 2003 Feb 15;97(4):934-59. doi: 10.1002/cncr.11105. PMID 12569593
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0193.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 68Gallium DOTATATE Imaging
Started | 341
Completed | 281
Not Completed | 60
Not completed — Withdrawal by Subject | 52
Not completed — Refuse treatment | 2
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 341
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 238
  >=65 years | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.89 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 147
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Black or African American | 24
  Native Hawaiian or Other Pacific Islander | 1
  Other | 7
  Race Unknown | 9
  White | 290
  Hispanic or Latino | 17
  Not Hispanic or Latino | 323
  Ethnicity Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 341

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions Detected Using the 68Gallium-DOTATATE Positron Emission Tomography (PET/Computed Tomography (CT)) Scan
Description: Patients with neuroendocrine tumors (NETs) were scanned with the 68Gallium-DOTATATE Positron Emission Tomography (PET/Computed Tomography (CT)) and the number of lesions detected are collected.
Time Frame: During PET Scan, up to 2 hours annually for up to 5 years
Population: Analysis was performed in the initial 131/341 participants scanned because 52 withdrew consent and 2 refused treatment. Subsequent scans in the remaining 156 participants were used to assess secondary objectives.
Measure: Number; unit: Number of lesions
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 131
Number of lesions | 847

2. Secondary Outcome: Mean Radiation Activity Between Low Grade and Intermediate Grade Neuroendocrine Tumor
Description: The radioactivity was assessed using intraoperative radiation detector following the 68Gallium-DOTATATE injection. Low grade neuroendocrine tumors is defined as tumors with slow cell division determined in histology. Low grade tumors is associated with the best outcome. Intermediate grade tumor is defined as the tumor with medium (3-20%) rate of actively dividing cells and is associated with less favorably outcome.
Time Frame: During radioguided surgery, up to 2 hours
Population: As of 12/22/14 when the analysis was performed, 14/140 subjects required surgical intervention with intraoperative radiation detector and thus were analyzed. 126 participants were not surgical candidates or did not receive intraoperative dose of 68Gallium-DOTATATE and did not have radiation detector.
Measure: Mean (Standard Deviation); unit: 511KeV count per ten seconds
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 14
511KeV count per ten seconds
  Low grade | 504.9 (534)
  Intermediate grade | 205 (147)

3. Secondary Outcome: Tumor Volume of Neuroendocrine Tumors Assessed by the 68Gallium-DOTATATE Scan
Description: Participants were scanned using the 68Gallium-DOTATATE Scan. Tumor volume more than 7ml is associated with shorter time to disease progression. Tumor volume more than 36 ml is associated with shorter disease specific survival.
Time Frame: During radioguided surgery, up to 2 hours
Population: 184/341 participants were analyzed because 52 withdrew consent and 2 refused treatment, 22 did not have a diagnosis of neuroendocrine tumor, and 81 had no 68Ga-DOTATATE uptake and were excluded.
Measure: Median (Full Range); unit: ml
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 184
ml | 9.24 [0.06 to 1136.7]

4. Secondary Outcome: Median Radioactivity of Tumors With High Expression of Somatostatin Receptor 2 Compared to Tumors With Intermediate Expression of Somatostatin Receptor 2
Description: High expression of somatostatin receptor 2 (SSTR2) is based on the intensity grading on immunohistochemistry. High SSTR2 expression may be associated with well-differentiated tumor and high avidity on DOTATATE scan, compared to intermediate or low expression of SSTR that can be seen in poorly differentiated and often aggressive neuroendocrine tumors. Because the correlation can only be from the comparison of preoperative DOTATATE and the tumors that were removed, it is a one time analysis. Subsequent DOTATATE studies are for surveillance and follow up for disease progression or recurrence.
Time Frame: During PET Scan, up to 2 hours annually
Population: As of 12/22/14 when the analysis was performed, 12/140 subj. required surgical intervention with intraoperative radiation detector & thus were analyzed. 12 subj. had their tumors analyzed for the expression of SSTR, 126 subj. were not surgical candidates or did not receive intraoperative dose of 68Gallium-DOTATATE & did not have radiation detector.
Measure: Median (Full Range); unit: Tumor to background ratio
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 12
Tumor to background ratio
  High expression | 6.5 [3.4 to 14.9]
  Low expression | 3.7 [3.5 to 6.3]
Statistical Analysis 1: Comparison: 68Gallium DOTATATE Imaging; Test type: Superiority; p = 0.23, Mann-Whitney

5. Secondary Outcome: The Number of Tumors Identified in Participants by the Radiation Detector During Radio-guided Surgery Using 68Gallium-DOTATATE
Description: Radio-guided surgery in neuroendocrine tumors using 68Gallium-DOTATATE was performed to detect tumors in the stomach and small bowel neuroendocrine tumors, pancreas, metastatic sites to lymph nodes and liver, and pheochromocytoma or paraganglioma. The number of tumors identified by the radiation detector were assessed.
Time Frame: Radio-guided surgery, up to 2 hours
Population: As of 02.14.2018 when the analysis was performed, 44/326 subjects required surgical intervention with intraoperative radiation detector and thus were analyzed for the number of tumors identified. 282 participants were not surgical candidates and did not receive intraoperative dose of 68 Gallium-DOTATATE and did not have radiation detector used.
Measure: Number; unit: Number of tumors
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 44
Number of tumors
  Stomach and small bowel | 23
  Pancreas tumors | 24
  Pheochromocytoma and paraganglioma | 6
  Liver metastasis | 9
  Metastatic lymph nodes | 71

6. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 50 months and 17 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 68Gallium DOTATATE Imaging
Number analyzed (Participants) | 341
Participants | 21

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 50 months and 17 days.
Arm/Group | 68Gallium DOTATATE Imaging
All-Cause Mortality (participants affected / at risk) | 16/341
Serious Adverse Events (participants affected / at risk) | 20/341
Other Adverse Events (participants affected / at risk) | 1/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Gallium DOTATATE Imaging (N=341)
Thromboembolic event (Vascular disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Death (unrelated to 68 Gallium DOTATATE) (General disorders) | 16 (16)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Gallium DOTATATE Imaging (N=341)
Alteration of consciousness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT01967537/Prot_SAP_ICF_000.pdf